CLINICAL TRIAL: NCT01182246
Title: Safety, Pharmacokinetics and Efficacy of AXP107-11 in Combination With Standard Gemcitabine (Gemzar®) Treatment in Patients With Locally Advanced or Metastatic, Unresectable, Adenocarcinoma of the Pancreas, Stage III-IV: A Prospective, Open Label, Multi-centre, Sequential Phase Ib/IIa Study
Brief Title: AXP107-11 in Combination With Standard Gemcitabine (Gemzar® ) Therapy for Treatment in Patients With Pancreatic Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Axcentua Pharmaceuticals AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AXP-CT-001
Record Dates: First submitted 2010-08-04; First posted 2010-08-16 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Adenocarcinoma
Keywords: adenocarcinoma; Pancreatic cancer
MeSH Terms: conditions — Adenocarcinoma; Pancreatic Neoplasms | interventions — Genistein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AXP107-11 (Experimental)
  Interventions: Drug: AXP107-11

INTERVENTIONS:
Drug: AXP107-11 — The drug substance, AXP107-11, is a crystalline form of genistein, a substance shown in literature data to target pancreatic tumor cells and also the tumor microenvironment and thus sensitizes tumors to chemotherapy. AXP107-11 is formulated in a capsule containing 2x100 mg of active substance.
  A maximum of four cohorts of three to six patients each will be treated with escalating dose levels of AXP107-11 alone (two weeks) and in combination with gemcitabine (one week).
  AXP107-11 capsules will be ingested orally twice daily (morning and evening) each day of the treatment period. In phase Ib, AXP107-11 will be administered once daily on the first treatment day (morning), followed by twice daily administrations continuously throughout the treatment period. When a minimum of six patients have been treated and evaluated on the maintenance dose (phase 1b), additional patients will be included directly into phase IIa.
  Other Names: genistein

SUMMARY:
The purpose of this study is to assess the effect and safety of AXP107-11 alone, and in combination with gemcitabine standard therapy, in patients with advanced or metastatic cancer of the pancreas. The safety, pharmacokinetics and efficacy of AXP107-11 in these patients will also be studied.

DETAILED DESCRIPTION:
The annual incidence rate of pancreatic cancer is almost identical to the mortality rate. Despite a low incidence rate, pancreatic cancer is the fourth leading cause of cancer mortality in both men and women. Today is the only potentially curative option of these patients complete surgical resection. However, a majority of the patients (up to 80%) are not eligible for surgery for different reasons.

Today is gemcitabine the accepted first-line treatment for these patients. Recent advances in the management of pancreatic cancer suggest that gemcitabine may be improved by combining it with other anticancer drugs.

One attractive therapeutic option is genistein. Genistein appears to sensitize tumors to chemotherapy both by targeting the tumor cells and also by targeting components of the tumor microenvironment.

However, the limited bioavailability of genistein in its known crystalline form has led to difficulties in attaining adequate plasma concentration, resulting in limited application and dissemination in the clinical setting. To overcome this limitation, a novel crystalline form of genistein with improved pharmaceutical properties is being used. AXP107-11, a crystalline salt of genistein has improved physiochemical properties (solubility, dissolution rate, bioavailability) as compared to the known crystalline form of genistein.

In this study, AXP107-11, will be investigated alone and in combination with gemcitabine in patients with pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of signing the informed consent
2. Histologically confirmed adenocarcinoma of the pancreas
3. Metastatic or locally advanced, unresectable disease stage III-IV.
4. Measurable disease according to the international criteria proposed by the Response Evaluation Criteria in Solid tumors (RECIST) for target lesions
5. Karnofsky Performance Status ≥ 70 at study entry (Appendix 18.4).
6. Life expectancy of more than three months
7. Negative pregnancy test for female patients
8. For fertile women, willingness to perform double-barrier contraception during study and for four weeks after last treatment
9. Able and willing to sign the informed consent form

Exclusion Criteria:

1. Previous or ongoing severe supraventricular or ventricular arrhythmia
2. Previous or ongoing coagulation or bleeding disorder (PTT > 1.5 x ULN)
3. HIV infection
4. Known hypersensitivity to any component of the AXP107-11 formulation or gemcitabine
5. Previous or ongoing significant liver pathology (other than metastases) and/or liver function disorders
6. Previous or ongoing significant chronic renal dysfunction
7. Previous or ongoing malignancy other than pancreatic cancer < five years prior to enrolment, except basal cell carcinoma treated locally
8. Cardiovascular disease, New York Heart Association (NYHA) classification III or IV16
9. Severe pulmonary obstructive or restrictive disease
10. Acute or chronic inflammation (autoimmune or infectious)
11. Significant active/unstable non-malignant disease likely to interfere with study assessments
12. Laboratory tests (hematology, chemistry) outside specified limits:

    * WBC ≤ 3 x 10³/mm³
    * ANC ≤ 1.5 x 10³/mm³
    * Platelets ≤ 100.000/mm³
    * Hb ≤ 9.0 g/dl (≤ 5.6 mmol/l)
    * PT/PTT > 1.5 x ULN
    * Serum creatinine > 130 μmol/l) or clearance < 60 ml/min
    * AST and/or ALT > 3 x ULN with the exception of patients with liver metastasis (> 5 x ULN)
    * Alkaline phosphatase > 3 x ULN
    * Total bilirubin > 3 x ULN
13. Immunotherapy within six weeks prior to enrolment.
14. Any chemotherapeutical treatment for pancreatic adenocarcinoma before enrolment
15. Any radiotherapy for pancreatic adenocarcinoma before enrolment except for treatment of bone metastases if target lesions are not included in the irradiated field
16. Major surgery within four weeks prior to enrolment
17. Pregnant or nursing woman
18. Participations in other interventional clinical study within four weeks of enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2010-11; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Determine the safety profile and the maximum tolerated dose (MTD) of AXP107-11 alone and when given in combination with gemcitabine standard therapy. | up to 6 months
  Safety (AEs, dose limiting toxicity, laboratory tests, vital signs, weight and ECG). MTD is defined at day 8.
To assess the effect of a combination therapy of AXP107-11 and gemcitabine on objective response rate defined as the percentage of patients who showed complete response (CR) or partial response (PR). | up to 6 months
  The tumour response evaluation will be performed according to RECIST (www.recist.org)

SECONDARY OUTCOMES:
To determine the pharmacokinetic (PK) profile of escalating doses of AXP107-11. | Day -13, 1, 8 and 15
  Plasma concentration of AXP107-11
To assess the safety and tolerability of a combination therapy of AXP107-11 and gemcitabine. | up to 6 months
  Assessed by occurrence of adverse events, abnormal changes in laboratory parameters, vital signs, ECG, relevant patient withdrawal and percentage of patients having reduction, omission or discontinuation of any study medication.
  Note: This is a secondary outcome measurement for patients in the phase IIa part of the study. This is a primary objective in phase Ib.
To assess the effect of a combination therapy of AXP107-11 and gemcitabine on overall survival (OS). | up to 6 months
To assess the effect of a combination therapy of AXP107-11 and gemcitabine on overall survival rate at six months after start of combination therapy. | up to 6 months
To assess the effect of a combination therapy of AXP107-11 and gemcitabine on time to progression (TTP). | up to 6 months
To assess the effect of a combination therapy of AXP107-11 and gemcitabine on palliation, defined as the percentage of patients who showed CR, PR or stable disease (SD). | up to 6 months
  The tumour response evaluation will be performed according to RECIST (www.recist.org)
To assess the effect of a combination therapy of AXP107-11 and gemcitabine on clinical benefit response, a composite of measurements of pain (pain intensity and analgesics consumption), Karnofsky performance status and weight. | up to 6 months
To assess the effect of combination therapy of AXP107-11 and gemcitabine on the tumor mass using F-18 fluorodeoxyglucose positron emission tomography (FDG-PET). | up to 6 months
  Will be performed on the first 5 patients in the phase IIa part of the study.
To assess the effect of a combination therapy of AXP107-11 and gemcitabine on symptom distress score as measured by the Edmonton Symptom Assessment System (ESAS). | up to 6 months
To assess the effect of a combination therapy of AXP107-11 and gemcitabine on quality of life as assessed by the EORTC QLQ-C30 questionnaire and the PAN26 module. | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Löhr, MD,PhD, Prof., Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Dept. of Clinical Science, Intervention and Technology, Div. of surgery, Karolinska University Hospital, Huddinge, Stockholm
  - Dept. of Oncology-Pathology, Karolinska University Hospital, Solna, Stockholm